CLINICAL TRIAL: NCT06921746
Title: Changes in the Urinary Microbiome and Metabolome During Treatment of the Overactive Bladder in Female Patients
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: University Hospital Bulovka (Unknown); Thomayer University Hospital (Other); Institute of Microbiology of the Czech Academy of Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: MicrOAB-001
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder; Urinary Microbiome; Urinary Metabolome
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overactive Bladder Patients: Patients with the symptoms of overactive bladder will be enrolled in this study group
  Interventions: Diagnostic Test: Urine Microbiological and Metabolomic Analysis

INTERVENTIONS:
Diagnostic Test: Urine Microbiological and Metabolomic Analysis — Microbiological and metabolomic analysis of a urine sample will be performed in the study subjects, before and after the end of the treatment.

SUMMARY:
This is a non-interventional study that will not pose any burden for the participants. The study subjects will be examined and treated in a standard manner according to current clinical recommendations for the treatment of overactive bladder (OAB). A portion of urine samples, which are routinely collected for biochemical and culture examinations as part of the diagnostic process, will be sent for examination of the characteristics of the urinary microbiome and metabolome (UMM) before and after treatment.

DETAILED DESCRIPTION:
Participation in the study will be offered to female patients who seek treatment for OAB symptoms themselves or are referred to centers participating in the project if a clinical diagnosis of idiopathic OAB is established in their case as part of the standard examination process.

Patients will be approached by one of the authorized team members with information about the possibility of participating in this study. If the patient is interested in participating in the study, she will give written informed consent to participate in the study. Subsequently, the inclusion and exclusion criteria for participation in the study will be verified and a standardized urine collection will be performed to examine the characteristics of UMM. At the same time, the patient will fill in standard questionnaires used to determine the severity of OAB symptoms.

To research changes in UMM during OAB treatment, patients will be divided into a group with a good treatment response (responders) and a group without a good treatment response (non-responders). The primary indicator of a good treatment effect (definition of responder) is a reduction in the number of episodes of severe urgency with or without urge incontinence over 3 days documented by a voiding diary by more than 50% compared to the state before treatment. Based on the available data, treatment success is anticipated in 60% of patients.

Subsequently, the study participants will be treated with standard drug treatment for five weeks. They will then be invited to evaluate the effect of treatment using standard symptom questionnaires. At the same time, a control standardized urine collection will be performed to examine the characteristics of UMM. The patients will then end their participation in the study and will continue their treatment according to the valid clinical recommendations for treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult women over 18 years of age
* Written consent to participate in the study
* Willingness to undergo OAB evaluation and treatment according to the protocol
* OAB symptoms lasting longer than 3 months
* At least 3 episodes of severe urgency with or without urge incontinence within 3 days documented by voiding diary
* OAB symptom score V8 questionnaire ≥ 8

Exclusion Criteria:

* Known congenital developmental defects of the urinary tract (congenital hydronephrosis, vesicoureteral reflux, renal agenesis and hypoplasia, multicystic and polycystic kidneys)
* Any previous treatment for OAB
* Recurrent urinary tract infections (more than 3 episodes in the last 12 months)
* Presence of a foreign body in the urinary tract - urolithiasis, urinary catheter, ureteral stent
* Acute or chronic diseases with possible influence on the function of the lower urinary tract (LUT)
* Rheumatoid arthritis
* Diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult women with symptoms of overactive bladder persisting longer than three months willing to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders to the OAB treatment | 6 weeks
  The proportion of study subjects responding to the treatment of OAB symptoms will be observed.

SECONDARY OUTCOMES:
Change in UMM characteristics between both groups | 6 weeks
  Changes in UMM characteristics based on laboratory examination will be compared between the two study groups (responders vs non-responders)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Krhut, prof., MD, PhD, Principal Investigator — University Hospital Ostrava
Locations (4):
- Czechia (4):
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - Thomayer University Hospital, Prague
  - Institute of Microbiology of the Czech Academy of Sciences, Prague
  - University Hospital Bulovka, Prague

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Nambiar AK, Arlandis S, Bo K, Cobussen-Boekhorst H, Costantini E, de Heide M, Farag F, Groen J, Karavitakis M, Lapitan MC, Manso M, Arteaga SM, Riogh ANA, O'Connor E, Omar MI, Peyronnet B, Phe V, Sakalis VI, Sihra N, Tzelves L, van Poelgeest-Pomfret ML, van den Bos TWL, van der Vaart H, Harding CK. European Association of Urology Guidelines on the Diagnosis and Management of Female Non-neurogenic Lower Urinary Tract Symptoms. Part 1: Diagnostics, Overactive Bladder, Stress Urinary Incontinence, and Mixed Urinary Incontinence. Eur Urol. 2022 Jul;82(1):49-59. doi: 10.1016/j.eururo.2022.01.045. Epub 2022 Feb 23. PMID 35216856
- [Background] Peyronnet B, Mironska E, Chapple C, Cardozo L, Oelke M, Dmochowski R, Amarenco G, Game X, Kirby R, Van Der Aa F, Cornu JN. A Comprehensive Review of Overactive Bladder Pathophysiology: On the Way to Tailored Treatment. Eur Urol. 2019 Jun;75(6):988-1000. doi: 10.1016/j.eururo.2019.02.038. Epub 2019 Mar 26. PMID 30922690
- [Background] Milsom I, Abrams P, Cardozo L, Roberts RG, Thuroff J, Wein AJ. How widespread are the symptoms of an overactive bladder and how are they managed? A population-based prevalence study. BJU Int. 2001 Jun;87(9):760-6. doi: 10.1046/j.1464-410x.2001.02228.x. PMID 11412210
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Agarwal A, Eryuzlu LN, Cartwright R, Thorlund K, Tammela TL, Guyatt GH, Auvinen A, Tikkinen KA. What is the most bothersome lower urinary tract symptom? Individual- and population-level perspectives for both men and women. Eur Urol. 2014 Jun;65(6):1211-7. doi: 10.1016/j.eururo.2014.01.019. Epub 2014 Jan 24. PMID 24486308
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-committee of the International Continence Society. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Neurourol Urodyn. 2002;21(2):167-78. doi: 10.1002/nau.10052. No abstract available. PMID 11857671
- [Background] Zheng H, Wang C, Yu X, Zheng W, An Y, Zhang J, Zhang Y, Wang G, Qi M, Lin H, Wang F. The Role of Metabolomics and Microbiology in Urinary Tract Infection. Int J Mol Sci. 2024 Mar 8;25(6):3134. doi: 10.3390/ijms25063134. PMID 38542107
- [Background] Gupta A, Dwivedi M, Mahdi AA, Gowda GA, Khetrapal CL, Bhandari M. 1H-nuclear magnetic resonance spectroscopy for identifying and quantifying common uropathogens: a metabolic approach to the urinary tract infection. BJU Int. 2009 Jul;104(2):236-44. doi: 10.1111/j.1464-410X.2009.08448.x. Epub 2009 Feb 23. PMID 19239442
- [Background] Bouatra S, Aziat F, Mandal R, Guo AC, Wilson MR, Knox C, Bjorndahl TC, Krishnamurthy R, Saleem F, Liu P, Dame ZT, Poelzer J, Huynh J, Yallou FS, Psychogios N, Dong E, Bogumil R, Roehring C, Wishart DS. The human urine metabolome. PLoS One. 2013 Sep 4;8(9):e73076. doi: 10.1371/journal.pone.0073076. eCollection 2013. PMID 24023812
- [Background] Colella M, Topi S, Palmirotta R, D'Agostino D, Charitos IA, Lovero R, Santacroce L. An Overview of the Microbiota of the Human Urinary Tract in Health and Disease: Current Issues and Perspectives. Life (Basel). 2023 Jun 30;13(7):1486. doi: 10.3390/life13071486. PMID 37511861
- [Background] Antunes-Lopes T, Vale L, Coelho AM, Silva C, Rieken M, Geavlete B, Rashid T, Rahnama'i SM, Cornu JN, Marcelissen T; EAU Young Academic Urologists (YAU) Functional Urology Working Group. The Role of Urinary Microbiota in Lower Urinary Tract Dysfunction: A Systematic Review. Eur Urol Focus. 2020 Mar 15;6(2):361-369. doi: 10.1016/j.euf.2018.09.011. Epub 2018 Sep 28. PMID 30270128
- [Background] Nelson DE, Dong Q, Van der Pol B, Toh E, Fan B, Katz BP, Mi D, Rong R, Weinstock GM, Sodergren E, Fortenberry JD. Bacterial communities of the coronal sulcus and distal urethra of adolescent males. PLoS One. 2012;7(5):e36298. doi: 10.1371/journal.pone.0036298. Epub 2012 May 11. PMID 22606251
- [Background] Salabura A, Luniewski A, Kucharska M, Myszak D, Dolegowska B, Ciechanowski K, Kedzierska-Kapuza K, Wojciuk B. Urinary Tract Virome as an Urgent Target for Metagenomics. Life (Basel). 2021 Nov 19;11(11):1264. doi: 10.3390/life11111264. PMID 34833140
- [Background] Morand A, Cornu F, Dufour JC, Tsimaratos M, Lagier JC, Raoult D. Human Bacterial Repertoire of the Urinary Tract: a Potential Paradigm Shift. J Clin Microbiol. 2019 Feb 27;57(3):e00675-18. doi: 10.1128/JCM.00675-18. Print 2019 Mar. PMID 30404941
- [Background] Mueller ER, Wolfe AJ, Brubaker L. Female urinary microbiota. Curr Opin Urol. 2017 May;27(3):282-286. doi: 10.1097/MOU.0000000000000396. PMID 28234750
- [Background] Monsen T, Ryden P. Flow cytometry analysis using sysmex UF-1000i classifies uropathogens based on bacterial, leukocyte, and erythrocyte counts in urine specimens among patients with urinary tract infections. J Clin Microbiol. 2015 Feb;53(2):539-45. doi: 10.1128/JCM.01974-14. Epub 2014 Dec 3. PMID 25472486
- [Background] Turnbaugh PJ, Ley RE, Hamady M, Fraser-Liggett CM, Knight R, Gordon JI. The human microbiome project. Nature. 2007 Oct 18;449(7164):804-10. doi: 10.1038/nature06244. PMID 17943116
- [Background] Cho I, Blaser MJ. The human microbiome: at the interface of health and disease. Nat Rev Genet. 2012 Mar 13;13(4):260-70. doi: 10.1038/nrg3182. PMID 22411464